CLINICAL TRIAL: NCT00568815
Title: Phase II Study of Rituximab Combined With ESHAP in Patients With Relapse or Refractory DLBCL
Brief Title: Rituximab Combined With ESHAP in Patients With Relapse or Refractory Diffuse Large B Cell Lymphoma (DLBCL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ye Guo, Dr., Fudan University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESHAP-DLBCL
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Lymphoma
Keywords: DLBCL; Rituximab; ESHAP; Efficacy; Toxicity
MeSH Terms: conditions — Lymphoma | interventions — ESAP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chemo (Experimental)
  Interventions: Drug: Rituximab combined with ESHAP

INTERVENTIONS:
Drug: Rituximab combined with ESHAP — Rituximab 375mg/m2 d1, VP-16 40mg/m2 d1-4, Ara-C 2g/m2 d5, DDP 25mg/m2 d1-4, Met 500mg/m2 d1-5
  Other Names: R-ESHAP

SUMMARY:
The purpose of this study is to evaluate the efficacy and toxicity of Rituximab combined with ESHAP (etoposide, methylprednisolone, cytarabine, and cisplatin) in the patients with diffuse large B cell lymphoma (DLBCL).

DETAILED DESCRIPTION:
The salvage therapy in the patients with DLBCL is still controversial. The investigators conducted this study to evaluate the efficacy and tolerability of Rituximab combined with ESHAP in the patients with DLBCL. The patients enrolled were defined to be relapsed or refractory after the first-line chemotherapy like CHOP or other CHOP-like regimens.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-70 years old
* Histological confirmed diffuse large B cell lymphoma
* ECOG performance status no more than 2
* Life expectancy of more than 3 months
* Relapse or refractory after the first-line chemotherapy of DLBCL
* No evidence of bone marrow involvement
* Normal laboratory values: hemoglobin > 8.0g/dl, neutrophil > 1.5×109/L, platelet > 80×109/L, serum creatine < 1× upper limitation of normal(ULN), serum bilirubin < 1× ULN, ALT and AST < 1.5× ULN

Exclusion Criteria:

* Pregnant or lactating women
* Serious uncontrolled diseases and intercurrent infection
* The evidence of CNS metastasis and bone marrow involvement
* History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* History of allergic reaction/hypersensitivity to rituximab

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Response rate | 6 weeks

SECONDARY OUTCOMES:
Toxicities | every cycle

CONTACTS AND LOCATIONS:
Overall Officials: Biyun Wang, M.D., Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China